CLINICAL TRIAL: NCT01759797
Title: Safety of Intravenous Transplantation of Bone Marrow Derived Mesenchymal Stem Cell in Patients With ALS
Brief Title: Intravenous Transplantation of Mesenchymal Stem Cell in Patients With ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Nerve-005
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2012-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS bone marrow mesenchymal stem cell intravenous injection
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell reciepient (Experimental): the patients with ALS who underwent intravenous injection of mesenchymal stem cell.
  Interventions: Biological: intra venous injection of stem cell

INTERVENTIONS:
Biological: intra venous injection of stem cell — Intra venous injection of mesenchymal stem cell
  Other Names: Stem cell transplantation

SUMMARY:
ALS is a debilitating disease with varied etiology characterized by rapidly progressive weakness, muscle atrophy and fasciculations, muscle spasticity, difficulty speaking (dysarthria), difficulty swallowing (dysphagia), and difficulty breathing (dyspnea). ALS is the most common of the five motor neuron diseases.Riluzole (Rilutek) is the only treatment that has been found to improve survival but only to a modest extent. It lengthens survival by several months, and may have a greater survival benefit for those with a bulbar onset. It also extends the time before a person needs ventilation support.Stem cell transplantation is a new hopeful way to improve the patients conditions and reduce the period of disabilities.

DETAILED DESCRIPTION:
In this study our purpose is to evaluate the safety of intraventricular injection of bone marrow derived mesenchymal stem cell.the patients who are eligible,underwent bone marrow aspiration.after cell separation and preparation,the patients underwent mesenchymal stem cell intraventricular injection by stereotaxis.after injection he will be under observed in ICU to monitor the adverse events(allergic and neurological side effects).patients are followed 1th,3th ,6th and 12 months after injection and each time these parameters are checked:ALS-FRS,EMG-NCV,FVC,side effect check list.

ELIGIBILITY:
Inclusion Criteria:

* - Age:18-65
* both gender
* duration of disease<2 years
* FVC>40% ALS-FRS>26

Exclusion Criteria:

* - neurological and psychiatric concomitant disease
* concomitant systemic disease
* treatment with corticosteroid,Ig,immunosuppressive during 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Fever | 48hours
  Evaluation the rate of fever 48 hours after cell transplantation
Unconsciousness | 48hours
  Evaluation the rate of unconsciousness 48hours after cell transplantation.
vomiting | 48hours
  Evaluation the rate of vomiting 48hours after cell transplantation.

SECONDARY OUTCOMES:
ALS-FRS | 6months
  Evaluation the improvement of ALS-FRS during 6months after cell transplantation.
FVC | 6months
  Evaluation the improvement of FVC (spectrometry )in patients after cell transplantation.
EMG-NCV | 6months
  Evaluation the improvement of EMG-NCV during 6 months after cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan department of degenerative medicine,Head of Royan celltherapy center; Seyed Masoud Nabavi, MD, Study Director — Proffessor assistant of Shahed University
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Nabavi SM, Arab L, Jarooghi N, Bolurieh T, Abbasi F, Mardpour S, Azimyian V, Moeininia F, Maroufizadeh S, Sanjari L, Hosseini SE, Aghdami N. Safety, Feasibility of Intravenous and Intrathecal Injection of Autologous Bone Marrow Derived Mesenchymal Stromal Cells in Patients with Amyotrophic Lateral Sclerosis: An Open Label Phase I Clinical Trial. Cell J. 2019 Jan;20(4):592-598. doi: 10.22074/cellj.2019.5370. Epub 2018 Aug 1. PMID 30124008
- See also: Related Info — http://Royaninstitute.org